CLINICAL TRIAL: NCT04469088
Title: Effectiveness of Dry Needling vs Manual Therapy in Patients With Temporomandibular Joint Disorders. A Randomized Controlled Trial.
Brief Title: Effectiveness of Dry Needling vs Manual Therapy in Patients With Temporomandibular Joint Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, María Catalina Osuna Pérez, Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUN.20/4.PRY
Record Dates: First submitted 2020-07-04; First posted 2020-07-13 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Joint Disorders; Dry Needling; Musculoskeletal Manipulations
Keywords: Temporomandibular joint disorders; Dry Needling; Manual Therapy; Orofacial disability; Neck Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental)
  Interventions: Other: Dry needling
- Manual Therapy Treatment (Active Comparator)
  Interventions: Other: Manual Therapy Treatment

INTERVENTIONS:
Other: Dry needling — Twenty-three patients with TJD will be allocated in Dry Needling Group. They will receive 3 sessions of dry needling separated for 4 days. This treatment will consist of puncturing the active myofascial trigger points (PGM) of the aforementioned muscles. Sterile acupuncture needles of 0.26 mm in diameter by 40 mm in length, guided with a plastic cannula of the Ener-qi brand, will be used. The area will be cleaned with alcohol and a deep puncture of the PGM will be performed, triggering local spasm responses. Needle through the muscle following the technique described by Hong (Hong et al. 1994). After the procedure, the area is compressed with cotton for 90 seconds.
  Arms: Dry Needling Group
Other: Manual Therapy Treatment — Twenty-three patients will be allocated in Manual Therapy (MT) Group for three sessions during 30 minutes. MT treatment will consist in the application of neuromuscular techniques of the temporal, masseter and sternocleidomastoid muscles and Jones techniques in the external pterygoid muscle. Neuromuscular techniques are performed with the index and major fingers to apply a transverse friction with enough pressure to feel vertical fibers of each muscle or produce a medium discomfort level. To perform the Jones technique on the external pterygoid muscle, the patient will be asked to open the mouth and deviate the jaw slightly towards the treated side in order to make room for the finger to be located between the upper jaw and the coronoid process. Once the trigger point is located, we press to trigger the pain and we look for neurological silence and we maintain the pressure for 90 seconds. Over time, we slowly withdraw the pressure and return to the position passively.
  Arms: Manual Therapy Treatment

SUMMARY:
Temporomandibular Joint Disorders (TJD) represent a set of conditions that involve pain and dysfunction of the temporomandibular joint. TJD are a frequent disability affection in the worldwide population and the 35% of affected present at least a symptom such as orofacial pain, mouth movement limitations and snapping or crying temporo-mandibular. Due to the increase of the incidence of the TJD the investigators propose to complete this study.

A randomized controlled trial with parallel groups have been designed and blind evaluation of the response variable.

The hypothesis is that dry needling produces a positive effect in the involved variables of this study in comparison with manual therapy.

The aim of this RCT is to compare the effectiviness of the application of manual therapy in comparison with dry needling in the perceived pain, mouth opening, the degree of cervical disability and the pressure-pain threshold (PPT) of myofascial trigger points (MTrP) in patiens with TJD.

ELIGIBILITY:
Inclusion Criteria:

Female and male subjects with an age of 18-65 years old with a TJD who meet at least two of the following inclusion criteria:

* Pain on palpation of the myofascial trigger points of the masseter, anterior temporal, posterior temporal, external pterygoid and sternocleidomastoid muscles (minimum 3 active trigger points).
* Pain in the temporomandibular joint.
* Limitation of mouth opening.
* Clicking of the temporomandibular joint.

Exclusion Criteria:

Subjects who present any of the following characteristics:

* fibromyalgia, orthodontia, systemic disease, syndrome or pathology with possible joint repercussions, patients undergoing treatment with NSAIDs, jaw fracture, mandibular surgery, non-collaborative patients or patients with phobia needles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At the beginning of treatment, the first day
  Pain Numeric Rating Scale to assess the intensity of the temporomandibular pain level in patients with TJD. Patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"),
Change from Baseline Pain intensity | At the ended of the first session, after an hour.
  Pain Numeric Rating Scale to assess the intensity of the temporomandibular pain level in patients with TJD. Patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"),
Change from Baseline Pain intensity | At the end of treatment, an average of 2 weeks.
  Pain Numeric Rating Scale to assess the intensity of the temporomandibular pain level in patients with TJD. Patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"),
Pain after trigger points pressure | At the beginning of treatment, the first day
  It will be measured by pressure algometry with the Wagner Force Ten model FDX algometer. Thus, a numerical value will be provided for the subjective perception of pain. The unit of measurement used is Kg / cm2. Once the trigger point is located within the taut band, pressure will be exerted perpendicular to the muscle plane and on the PGM through the support surface of the device. We increase the pressure at a constant rate of 1 kg / cm2 / s. When the pressure becomes a painful stimulus, the individual must raise his hand to warn us.
Change from Baseline Pain after trigger points pressure | At the ended of the first session, after an hour.
  It will be measured by pressure algometry with the Wagner Force Ten model FDX algometer. Thus, a numerical value will be provided for the subjective perception of pain. The unit of measurement used is Kg / cm2. Once the trigger point is located within the taut band, pressure will be exerted perpendicular to the muscle plane and on the PGM through the support surface of the device. We increase the pressure at a constant rate of 1 kg / cm2 / s. When the pressure becomes a painful stimulus, the individual must raise his hand to warn us.
Change from Baseline Pain after trigger points pressure | At the end of treatment, an average of 2 weeks
  It will be measured by pressure algometry with the Wagner Force Ten model FDX algometer. Thus, a numerical value will be provided for the subjective perception of pain. The unit of measurement used is Kg / cm2. Once the trigger point is located within the taut band, pressure will be exerted perpendicular to the muscle plane and on the PGM through the support surface of the device. We increase the pressure at a constant rate of 1 kg / cm2 / s. When the pressure becomes a painful stimulus, the individual must raise his hand to warn us.
Open mouth movements | At the beginning of treatment, the first day
  It will be measured with a validated ruler in centimeters.
Change from Baseline open mouth movements | At the ended of the first session, after an hour.
  It will be measured with a validated ruler in centimeters.
Change from Baseline open mouth movements | At the end of the tratment, an average of 2 weeks
  It will be measured with a validated ruler in centimeters.
Neck Disability Index | At the beginning of treatment, the first day.
  It will measured with the Spanish version of the Neck Disability Index. The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. Higher scores mean a worse outcome.
Change from Baseline Neck Disability Index | At the end of the treatment, an average of 2 weeks
  It will measured with the Spanish version of the Neck Disability Index. The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Demographic variables | At the beginning of the treatment, the first day.

CONTACTS AND LOCATIONS:
Overall Officials: María Catalina Osuna Pérez, PhD, Principal Investigator — University of Jaén
Locations (1):
- Clínica de Fisioterapia y Rehabilitación Miophys S.C.A., Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pessoa DR, Costa DR, Prianti BM, Costa DR, Delpasso CA, Arisawa EALS, Nicolau RA. Association of facial massage, dry needling, and laser therapy in Temporomandibular Disorder: case report. Codas. 2018 Nov 29;30(6):e20170265. doi: 10.1590/2317-1782/20182017265. PMID 30517267
- [Result] Blasco-Bonora PM, Martin-Pintado-Zugasti A. Effects of myofascial trigger point dry needling in patients with sleep bruxism and temporomandibular disorders: a prospective case series. Acupunct Med. 2017 Mar;35(1):69-74. doi: 10.1136/acupmed-2016-011102. Epub 2016 Oct 3. PMID 27697769
- [Result] Gonzalez-Perez LM, Infante-Cossio P, Granados-Nunez M, Urresti-Lopez FJ, Lopez-Martos R, Ruiz-Canela-Mendez P. Deep dry needling of trigger points located in the lateral pterygoid muscle: Efficacy and safety of treatment for management of myofascial pain and temporomandibular dysfunction. Med Oral Patol Oral Cir Bucal. 2015 May 1;20(3):e326-33. doi: 10.4317/medoral.20384. PMID 25662558